CLINICAL TRIAL: NCT03286894
Title: AQUAPed: Validation Study of AQUA© Questionnaire Modified for Childhood
Acronym: AQUAPed
Status: Completed | Type: Observational
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, MD. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: 7/2017_D
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1264 healthy schoolchildren: There is only one study group consisting of 1264 children recruited at school.

SUMMARY:
The AQUA© questionnaire developed in 2008 is a validated tools for the screening of allergic diseases in adult athletes. The objective of the present study is to develop and validate a modified version of the AQUA© questionnaire to be used in childhood. In this phase, the validation is intended to assess the reliability of the information collected through the AQUA© modified version: question difficulty and response patterns with respect to children characteristics (in particular age, sex and physical activity). In particular, the focus will be on the "core questions", i.e. the indicators of allergic disorders. This is a cross-sectional study on 1264 healthy schoolchildren aged 8 to 14 years.

ELIGIBILITY:
Inclusion Criteria:

* Aforementioned sex and age criteria.

Exclusion Criteria:

* Respiratory infections in the previous 3 weeks;
* Immunological or metabolic systemic disease;
* Major malformations of the upper airways;
* Active smoker.

Ages: 8 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: The study population consists of 1264 healthy schoolchildren, both males and females, aged 8 to 14 years, recruited in 7 primary and secondary schools of the city of Palermo.
Sampling Method: Non-Probability Sample
Enrollment: 1264 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Question difficulty | Study end (4 months)
  Comprehensibility (or difficulty) of the questions, especially the "core questions", will be assessed by the percentages of non-response possibly stratified by children characteristics (in particular age, sex and physical activity).

SECONDARY OUTCOMES:
Patterns of missing response | Study end (4 months)
  Possible tendency to skip consecutive questions will be assessed by studying the association between the presence of missing (0 = answer missing, 1 = answer given) in sequence (tetrachoric correlation).
Patterns of non-missing responses | Study end (4 months)
  Analysis of the distribution of non-missing responses, possibly stratified by children characteristics (in particular age, sex and physical activity).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology (IBIM), National Research Council, Palermo, Sicily, Italy